CLINICAL TRIAL: NCT05748665
Title: Effect of Remimazolam Induction on the Recovery Quality After Day Surgery in Elderly Patients: a Comparison Study With Etomidate
Brief Title: Effect of Remimazolam on the Recovery Quality After Day Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY20222277-F-1
Record Dates: First submitted 2023-01-06; First posted 2023-03-01 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-01

CONDITIONS: Elderly Patients; Ambulatory Surgery
MeSH Terms: interventions — Etomidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remimazolam (Experimental): remimazolam induction
  Interventions: Drug: Remimazolam besylate
- etomidate (Active Comparator): etomidate induction
  Interventions: Drug: etomidate

INTERVENTIONS:
Drug: Remimazolam besylate — Using remimazolam for induction of general anesthesia
  Arms: remimazolam
Drug: etomidate — Using etomidate for induction of general anesthesia
  Arms: etomidate

SUMMARY:
The goal of this clinical trial is to compare remimazolam and etomidate in inducing quality of recovery after day surgery for laryngeal mask general anesthesia in elderly patients. The main question it aims to answer is:

• The quality of postoperative recovery induced by remimazolam for laryngeal mask general anesthesia in elderly patients undergoing day surgery is not inferior to that induced by etomidate Participants will be given remimazolam to induce anesthesia。 Researchers will compare etomidate to see if the quality of postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* undergoing day surgery under laryngeal mask anesthesia
* American society of anesthesiologists (ASA) grade 1-3
* BMI<30kg/m2

Exclusion Criteria:

* have benzodiazepines drugs in the latest month cognitive dysfunction
* Cognitive dysfunction and neuropsychiatric disorders
* It was estimated as a difficult airway
* There was a history of adrenal insufficiency, porphyria, or chronic corticosteroid therapy
* There is a contraindication or allergy to benzodiazepines, opioids, etomidate and its components

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
The quality of recovery 15 | postoperative day 1
  The main goal of this study was to assess the QoR using the QoR-15 questionnaire, which is a global measure of recovery after surgery that evaluates five dimensions of recovery: physical comfort (5 items), physical independence (2 items), emotional state (4 items), psychological support (2 items), and pain (2 items). Each item is rated on an 11- point scale based on its frequency on the questionnaire (greater score at greater frequency for positive items and less frequency for negative items). The total score ranged from 0 (poorest recovery quality) to 150 (best recovery quality).

SECONDARY OUTCOMES:
The time of loss of consciousness | within 3 minutes after the end of the intravenous anesthetic
  The time of disappearance of the eyelash reflex within 3 minutes after the end of the intravenous anesthetic
Adverse events | During stay of post anesthesia care unit (up to 30minutes）
  Respiratory, cardiovascular and neurological system adverse events
the mean blood pressure，the systolic blood pressure ，the diastolic pressure | From 5 minutes before anesthesia induction to the time point surgery start
  Vital signs at different time points
heart rate | From 5 minutes before anesthesia induction to the time point surgery start
  heart rate at different time points
pulse oxygen saturation | From 5 minutes before anesthesia induction to the time point surgery start
  pulse oxygen saturation at different time points

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Fourth military medical university, Xijing Hospital, Xi'an, Shannxi
  - Xi 'an International Medical Center Hospital, Xi'an, Shannxi
  - Yan 'an University Affiliated Hospital, Yanan, Shannxi

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT05748665/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT05748665/ICF_001.pdf